CLINICAL TRIAL: NCT04694703
Title: Changing of Trace Element, Homocysteine, Oxidative Stress Parameters and Physical Activity Levels in Patients Diagnosed With COVID-19 Before and After COVID-19 Treatment
Brief Title: Changing of Trace Element, Homocysteine, Oxidative Stress Parameters and Physical Activity Levels in Covid-19
Status: Completed | Type: Observational
Sponsor: Izmir Bakircay University (Other)
Collaborators: Cigli Regional Training Hospital (Other); Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Kadirhan Ozdemir, PT, PhD., Assist. Prof., Izmir Bakircay University
Other Study IDs: 2020-12-142
Record Dates: First submitted 2021-01-03; First posted 2021-01-05 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Covid19
Keywords: Covid-19 (SARS-CoV-2); Trace element; Homocystein; Oxidative stress parameters; Physical activity level
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Covid-19 group: Patients diagnosed with COVID-19 will be enrolled in this group.
  Interventions: Drug: Covid-19 group

INTERVENTIONS:
Drug: Covid-19 group — Routine COVID-19 treatment

SUMMARY:
With the rapid spread of COVID-19 (SARS-CoV-2) disease all over the world and the announcement of a pandemic, researches on many different drug approaches have begun and these researches continue today. Considering the absence of a specific treatment for the disease yet and the urgency of the situation, drugs previously licensed for the treatment of other diseases and thought to be effective in COVID-19 have started to be used. Ongoing studies are conducted on the effectiveness, possible side effects and safety of these drugs in COVID-19, but there is no clear information yet. It is thought that the anti-inflammatory and antioxidant properties of some vitamins and trace elements may be associated with positive results in COVID-19 patients, and the physiological roles of these vitamins and trace elements in COVID 19 have been demonstrated by studies. It is important to investigate the levels of free radicals known to be effective in the development of cardiovascular disease due to homocysteine and oxidative stress, which can provide information on determining the risk of cardiovascular complications in the COVID-19 pandemic. In addition, as the decrease in physical activity levels of individuals in the COVID-19 pandemic may cause possible secondary complications such as an increase in the risk of cardiovascular disease, determining the physical activity levels of individuals and encouraging them to physical activity is another important parameter to minimize the negative effects of the process. It is thought that investigating the effects of the treatment approaches used in COVID-19 on trace element, homocysteine, oxidative stress parameters and physical activity levels will provide useful information in determining the factors underlying better clinical results. This study was planned to be carried out between 6-31 January 2021 in order to compare the trace element, homocysteine, oxidative stress parameters and physical activity levels before and after treatment for COVID-19 disease in COVID-19 patients who applied to Izmir Bakircay University Cigli Training and Research Hospital (Cigli Regional Training Hospital) and hospitalized in the COVID-19 service. Research data will be obtained from blood samples taken from participants. In addition, data on physical activity levels will be collected through a questionnaire. After analyzing the data obtained from the research with appropriate statistical methods, the data will be evaluated.

DETAILED DESCRIPTION:
Since December 2019, the new severe acute respiratory syndrome coronavirus 2, called SARS-CoV-2, has spread rapidly to almost every country that causes coronavirus disease-19 (COVID-19) pneumonia. Currently, there is no specific treatment for COVID-19 with proven safety and effectiveness. In order to find an effective treatment for this disease, more than 100 randomized controlled trials are currently being conducted with many drugs, some of them are expected to be announced in the coming months. It is known that the use of treatment options within the framework of randomized controlled studies and based on information obtained from other scientific studies is more rational. However, due to the urgency of the current situation and the limited scientific data, treatment options with limited data on their effectiveness are widely used for these patients all over the world. As in general of viral infections, the data obtained from SARS and influenza suggest that early initiation of antiviral treatment is more beneficial, and antiviral drugs should be started as early as possible. The combined use of possible treatment options in COVID-19 patients should be considered on a patient-specific basis and by evaluating all the relevant literature, and attention should be paid to the interactions and adverse effects of the drugs used.

Since it will take a long time to find a treatment specific to COVID-19, during the current pandemic, drugs such as hydroxychloroquine, favipiravir, remdesivir, lopinavir-ritonavir, which have been previously licensed for the treatment of other diseases in humans, have been widely used in these indications, have been shown to be safe and are effective in SARS CoV-2 in vitro, have been recommended and used. Numerous studies are still ongoing on the efficacy and safety of these drugs in COVID-19.

The clinical picture of COVID-19 can be heterogeneous, ranging from asymptomatic to severe disease, which can be associated with a cytokine storm. The pathogenesis of COVID-19 is not fully understood, but is likely multifactorial and, in severe cases, with a systemic hyperinflammatory response and associated thromboembolic complications.

It may be beneficial for patients infected with COVID-19 due to the anti-inflammatory and antioxidant properties of certain vitamins and nutrients. Vitamins such as A, B, C, D, E and folate and trace elements such as iron, zinc, magnesium, selenium and copper play important roles in supporting both innate and adaptive immune systems.

High plasma homocysteine levels significantly increase the incidence of vascular damage in both small and large vessels. Concentrations above the 90th percentile are associated with an increased risk of degenerative and atherosclerotic processes in the coronary, cerebral and peripheral circulatory systems. Although homocysteine is an effective cardiovascular risk biomarker and is critical for cardiovascular complications in hospitalized COVID-19 patients, studies on this parameter have not focused much on laboratory markers useful for clinical evaluation of COVID-19.

Free radicals are continuously formed at the active site of enzymes as intermediates in enzymatic reactions occurring during cell metabolism. Reactive oxygen species and reactive nitrogen, known as intermediates, sometimes leach from the active site of enzymes and accidentally interact with molecular oxygen and form free oxygen radicals. Lipids, proteins, enzymes, carbohydrates, and DNA can be damaged due to oxidative stress, random breaks and bonds in DNA chains may occur as a result of damage to membranes, damage to enzymes and structural proteins may result in cell death, and these phenomena constitute the molecular basis in the development of cancer, neurodegenerative and cardiovascular diseases, diabetes and autoimmune disorders.

The general recommendation for thinking that an adult is physically active is to achieve at least 150 minutes of moderate or 75 minutes of vigorous vigorous activity per week, or an equivalent combination of both, and involving sedentary behavior, energy expenditure ≤ 1.5 metabolic equivalent (MET), while lying down, leaning, It is defined as any waking behavior practiced while sitting or standing. As the disease spreads all over the world, healthy people are asked to stay at home for a long time. As a result, COVID-19 has radically changed the determinants of both behaviors (individual, interpersonal, environmental, regional or national policies and global). Accordingly, it can be said that regular and joint activities decrease due to isolation and limitations, especially in the first weeks when the population has limited chances to find alternatives to keep active even at home, and reducing sedentary behavior during closure poses a significant challenge. Because of this situation, physical activity in the home environment is strongly encouraged by public health advocates to prevent the potential harmful effects of protective lifestyle regulations due to COVID-19 and to prevent the restrictions from causing physical inactivity.

The purpose of this study is to compare the trace element, homocysteine, oxidative stress parameters and physical activity levels before and after COVID-19 treatment according to the COVID-19 treatment guide published by Ministry of Health, Republic of Turkey.

ELIGIBILITY:
Inclusion Criteria:

* To agree to participate in the study voluntarily,
* Having a diagnosis of COVID-19,

Exclusion Criteria:

* Having been taking trace element supplements for the last 2 weeks and/or currently,
* Patients who do not need hospitalization,
* Having a diagnosis of kidney failure and/or heart failure,
* Being pregnant,
* Body mass index over 40 kg/m2

Ages: 35 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants in Group I and Group II will be included the study from Izmir Bakircay University Cigli Training and Research Hospital (Cigli Regional Training Hospital).
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-08-29 (Actual)

PRIMARY OUTCOMES:
Change of the levels of Trace Element at baseline and discharge | At baseline and immediately before the discharge
  Serum trace elements (zinc, selenium, potassium, sodium, calcium, magnesium, copper) levels will be determined by venous blood samples taken from the participants. Serum trace element levels samples will be analyzed using the atomic absorption spectrophotometry (AAS) method.
Change of Physical Activity Level at baseline and discharge | At baseline and immediately before the discharge
  International Physical Activity Questionnaire will be used to determine the level of physical activity.
Change of the levels of Homocystein at baseline and discharge | At baseline and immediately before the discharge
  Homocystein levels will be studied by using Enzyme Chemiluminescence Immunoassay (ECLIA) in Medical Biochemistry Laboratory.
Change of the levels of Oxidative Stress Parameters at baseline and discharge | At baseline and immediately before the discharge
  Oxidative Stress Parameters including Superoxide Dismutase (SOD), Malondialdehyde (MDA), Total Antioxidant Level (TAL) / Total Oxidant Level (TOL) will be studied by photometric method in Medical Biochemistry Laboratory.

SECONDARY OUTCOMES:
Change of the levels of Routine Blood Samples (Hemogram) at baseline and discharge | At baseline and immediately before the discharge
  Hemogram results will be taken from patient files.
Change of the levels of Routine Blood Samples (vitamin D, Troponin T, D-Dimer, iron and ferritin) at baseline and discharge | At baseline and immediately before the discharge
  Levels of vitamin D, Troponin T, D-Dimer, iron and ferritin will be taken from patient files.
Change of the levels of Routine Blood Samples (C-reactive protein (CRP) and procalcitonin) at baseline and discharge | At baseline and immediately before the discharge
  Levels of C-reactive protein (CRP) and procalcitonin will be taken from patient files.
Change of the levels of Routine Blood Samples (uric acid, chlorine, blood urea nitrogen (BUN) creatine, albumin and bilirubin) at baseline and discharge | At baseline and immediately before the discharge
  Levels of uric acid, chlorine, blood urea nitrogen (BUN) creatine, albumin and bilirubin will be taken from patient files.

CONTACTS AND LOCATIONS:
Locations (1):
- Kadirhan Ozdemir, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Adult Patient Treatment Guide for COVID-19 (Ministry of Health, Republic of Turkey) — https://covid19.saglik.gov.tr/TR-66926/eriskin-hasta-tedavisi.html